CLINICAL TRIAL: NCT02037802
Title: Caudal Extradural Catheterization in Pediatric Renal Transplant: Effect on Perioperative Hemodynamics and Pain Scoring.
Brief Title: Caudal Epidural Catheterization in Pediatric Renal Transplant: Effect on Hemodynamics and Pain After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Mohamed Abd el moneim Soaida, MD, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SMS2014-1
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Renal Failure
Keywords: caudal; epidural; pediatric; renal; transplant; hemodynamics
MeSH Terms: conditions — Renal Insufficiency | interventions — Meperidine; Propofol; Bupivacaine; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- caudal epidural catheterization group (Active Comparator): 30 patients received continuous intra and post-operative caudal epidural infusion of bupivacaine 0.125% with fentanyl (2 microgram/ml) over 24 hours
  Interventions: Device: B-Braun, Perifix® ONE Paed, Germany; Drug: Pethidine; Drug: Propofol; Drug: Bupivacaine; Drug: Fentanyl
- control group (Sham Comparator): 30 patients didn't receive caudal epidural analgesia
  Interventions: Drug: Pethidine; Drug: Propofol; Drug: Fentanyl

INTERVENTIONS:
Device: B-Braun, Perifix® ONE Paed, Germany — caudal epidural catheterization bupivacaine fentanyl
  Arms: caudal epidural catheterization group
Drug: Pethidine — pethidine intravenous at a dose 1mg/kg when pain score more than 5 postoperative rescue analgesia
Drug: Propofol — fentanyl propofol atracurium besylate
Drug: Bupivacaine
  Arms: caudal epidural catheterization group
Drug: Fentanyl

SUMMARY:
pain control in pediatric renal transplant is a major concern. the main goal during anesthesia of renal transplant in pediatrics is to maintain hemodynamics in a range close to that of the adult donor. epidural analgesia is thought to be very effective in pain control. this study emphasises the ease of application of epidural catheter via the caudal route to the lower thoracic level; avoiding possible complications that may arise from lumbar or thoracic routes, and its effects on hemodynamics when using analgesic doses of local anesthetics and narcotics.

ELIGIBILITY:
Inclusion Criteria:

* 3-12 years
* end stage renal disease
* no known allergy to bupivacaine
* both sexes

Exclusion Criteria:

* known allergy to bupivacaine
* inflammation at caudal area
* spinal cord deformity

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood pressure | from the induction of anesthesia till end of surgery at half an hour intervals
  measure systolic and diastolic blood pressure

SECONDARY OUTCOMES:
postoperative blood pressure | from the time of transfer of the patient to the intensive care unit at one hour intervals for 24 hours
  record systolic and diastolic blood pressure every hour for the first 24 hours postoperative
intraoperative central venous pressure | fromom the induction of anesthesia till end of surgery at half an hour intervals
postoperative heart rate | from the time of transfer of the patient to the intensive care unit at one hour intervals for 24 hours
postoperative central venous pressure | from the time of transfer of the patient to the intensive care unit at one hour intervals for 24 hours
intraoperative heart rate | from the induction of anesthesia till end of surgery at half an hour intervals

OTHER OUTCOMES:
pain scoring system (objective behavioural pain score) | from the time of transfere to the nephrology ICU, every hour for the first 24 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Sherif M Soaida, M.D., Principal Investigator — Cairo University
Locations (1):
- Faculty of medicine, Cairo University, Cairo, Egypt

REFERENCES:
- [Derived] Soaida SM, ElSheemy MS, Shouman AM, Shoukry AI, Morsi HA, Salah DM, Fadel FI, Bazaraa HM. Caudal extradural catheterization in pediatric renal transplant and its effect on perioperative hemodynamics and pain scoring: a prospective randomized study. J Anesth. 2016 Feb;30(1):47-54. doi: 10.1007/s00540-015-2087-8. Epub 2015 Oct 22. PMID 26493396